CLINICAL TRIAL: NCT02597972
Title: Reverse Total Shoulder Arthroplasty Versus Open Reduction Internal Fixation of 3 &Amp; 4-Part Proximal Humerus Fractures: A Randomized Prospective Study
Brief Title: Reverse Total Shoulder Arthroplasty Versus Open Reduction Internal Fixation of 3&4 Part Proximal Humerus Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: project opened under new PI
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joaquin Sanchez-Sotelo, M.D., Ph.D., Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-004148
Record Dates: First submitted 2015-09-17; First posted 2015-11-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Closed Fracture Proximal Humerus, Four Part
MeSH Terms: interventions — Arthroplasty, Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Reduction Internal Fixation Proximal Humerus (Active Comparator): The patients randomized into the ORIF group will receive standard surgical treatment of their proximal humerus fracture with a proximal humeral locking plate.
  Interventions: Procedure: Fracture repair
- Reverse Total Shoulder Arthroplasty (Active Comparator): The patients randomized into the RTSA group will receive standard surgical treatment of their proximal humeral fracture with a Reverse Total Shoulder Arthroplasty.
  Interventions: Procedure: Fracture repair with joint replacement

INTERVENTIONS:
Procedure: Fracture repair
  Arms: Open Reduction Internal Fixation Proximal Humerus
Procedure: Fracture repair with joint replacement
  Arms: Reverse Total Shoulder Arthroplasty

SUMMARY:
Will patients who suffer complex humerus fractures have better functional outcomes and less implant failure with shoulder replacement (reverse total shoulder arthroplasty, RTSA) compared to shoulder repair (open reduction and internal fixation, ORIF)?

DETAILED DESCRIPTION:
The purpose of this study is to compare validated clinical and functional outcomes between patients who acutely present with 3 and 4-part proximal humerus fractures treated with either ORIF or RTSA.

ELIGIBILITY:
Inclusion

* Neer 3 and 4-part proximal humerus fractures.
* Age greater than and equal to 70 years old.
* Functional deltoid musculature (axillary nerve intact).

Exclusion

* Less than 70 years old.
* Dementia or inability to provide adequate follow up.
* Associated injuries: injuries of ipsilateral limb, complete brachial plexopathy, vascular injury and polytrauma.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
To measure the change using the chi-square tests for lowering the pain score of the patients | base line to 2 years
  threshold of statistical significance will be set at α = 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Sanchez-Sotelo, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials